CLINICAL TRIAL: NCT04147702
Title: Evaluation of Balance, Trunk Muscle Endurance and Pulmonary Functions in Dancers
Brief Title: Evaluation of Balance and Trunk Muscle Endurance in Dancers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ozden Ozkal, Principal Investigator, Hacettepe University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: GO 19/511
Record Dates: First submitted 2019-10-30; First posted 2019-11-01 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Balance; Distorted; Sports Injury
Keywords: Balance; Dancer; Respiratory muscle; Trunk muscle
MeSH Terms: conditions — Athletic Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group: Balance analysis (Experimental): fifty dancers will be evaluated in this study.Trunk muscle endurance, pulmonary functions and balance will be assessed.
  Interventions: Other: Balance analysis
- Control Group:Balance Analysis (Active Comparator): fifty healthy subjects will be evaluated in this study.Trunk muscle endurance, pulmonary functions and balance will be assessed.
  Interventions: Other: Balance analysis

INTERVENTIONS:
Other: Balance analysis — Balance analysis is assessment method to estimate deterioration of postural control.

SUMMARY:
This study evaluates endurance of trunk muscles, balance and pulmonary functions in dancers. The participants will be evaluated trunk muscles endurance, pulmonary functions and balance which evaluated by computerized force plate system.

DETAILED DESCRIPTION:
Dance is a form of exercise associated with movements that require balance, flexibility, endurance and skill. In addition to maintaining balance, the endurance of the trunk stabilizer muscles has an important role in sport-specific activities, coordination and athletic performance. Studies which conducted on dancers are mainly focused on abdominal muscle strength / endurance, lower extremity strength and physical performance. In the literature, it was reported that 40-84% of professional dancers and 26-51% of professional dancers had musculoskeletal injuries, particularly lower extremity problems. It is very important to regain balance after returning to the dance after foot and ankle injuries. Considering the function of the trunk as a bridge between the lower and upper extremities, it is known that trunk muscles play a fundamental role in regaining balance. However, in the literature, there is no study showing the effects of trunk stabilizer muscles (abdominal, dorsal extensor, lateral flexor and diaphragm), trunk flexibility and dance-specific properties on balance in dancers. As a result of this study, it is aimed to show the effect of dance on balance and related parameters and to reveal the factors affecting the balance.

ELIGIBILITY:
Inclusion Criteria:

* able and willing to complete the informed consent process.
* performing a sportive latin dancers as a competitive

Exclusion Criteria:

* having a pulmonary system disease
* having a cardiac system disease
* to do regular sports in addition to danc for the last three months

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Limits of Stability | 10 minutes
  Limits of stability test evaluates dynamic balance of participants. Computerized balance system measured limits of stability for forward, backward, right and left side movements. It calculates the maximum distance a person can lean without losing balance. The unit of measure is centimeters. The higher value is indicated the better balance
Postural sway | 10 minutes
  Postural sway in centimeters by computerized balance system

SECONDARY OUTCOMES:
Forced Vital Capacity | 15 minutes
  It is the total amount of air exhaled during the test. After three trial, the best forced vital capacity value is the outcome
Forced Expiratory Volume in 1 Second | 15 minutes
  Forced Expiratory Volume in 1 Second is the volume exhaled during the first second of a forced expiratory maneuver started from the level of total lung capacity. After three trial, the best FVC value is the outcome.
Forced Expiratory Volume in 1 Second / Forced Vital Capacity | 15 minutes
  The ratio of Forced Expiratory Volume in 1 Second / Forced Vital Capacity. This formule is calculated by measuring device. After three trial, the best value is the outcome
Maximal Inspiratory Pressure | 15 minutes
  It is a measure of the strength of inspiratory muscles, primarily the diaphragm. It is obtained by having the patient inhale as strongly as possible against a mouthpiece. After three trial, the best value is the outcome.
Maximal Expiratory Pressure | 15 minutes
  It is a measure of the strength of respiratory muscles, obtained by having the patient exhale as strongly as possible against a mouthpiece. After three trial, the best value is the outcome.
Peak Expiratory Flow | 15 minutes
  Peak Expiratory Flow is a person's maximum speed of expiration, as measured with a peak flow meter, a small, hand-held device used to monitor a person's ability to breathe out air. After three trial, the best value is the outcome.
forced expiratory flow | 15 minutes
  Forced expiratory flow is the flow (or speed) of air coming out of the lung during the middle portion of a forced expiration.
Trunk muscle endurance | 15 minutes
  The time to maintain the specified positions is recorded.
Trunk flexibility | 1 minutes
  To measure flexibility, the participant will be instructed to push the yardstick placed at the edge of the box while holding the legs straight and the hands parallel to the floor as far as she could. this test in centimeters by measuring tape.

CONTACTS AND LOCATIONS:
Locations (1):
- Ozden Ozkal, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No